CLINICAL TRIAL: NCT04377477
Title: Pilot Study on the Feasibility of Low Dose Radiotherapy for SARS-Cov-2 Pneumonitis (COVID-19 Low Dose Radiotherapy - COLOR 19)
Brief Title: COVID-19 Pneumonitis Low Dose Lung Radiotherapy (COLOR-19)
Acronym: COLOR-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Stefano Maria Magrini, Prof, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP 4097
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: COVID-19
Keywords: RADIOTHERAPY; PNEUMONITIS
MeSH Terms: conditions — COVID-19; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lung low dose radiotherapy (Experimental): Irradiation of the lungs, administered in a single fraction at the average prescription dose of 0.7 Gy
  Interventions: Radiation: Single fraction whole lung radiotherapy

INTERVENTIONS:
Radiation: Single fraction whole lung radiotherapy — Participants will undergo irradiation of the lungs, administered in a single fraction at the average prescription dose of 0.7 Gy

SUMMARY:
Low-dose radiotherapy treatment delivered to both lungs in patients with immune-related pneumonia following COVID-19 infection is backed up by biological and clinical bases that justify its use as a possible therapeutic option in these patients. This is a preliminary exploratory study (non-pharmacological interventional) to evaluate the feasibility and tolerability of low-dose radiotherapy treatment of SARS-Cov-2 immune-mediated pneumonia, for the subsequent implementation of a phase II study.This is a preliminary, monocentric, single-arm, interventional, non-pharmacological exploratory study. All enrolled patients will be treated with low-dose radiotherapy. Participants will undergo irradiation of the lungs, administered in a single fraction at the average prescription dose of 0.7 Gy (further details in the dedicated section).

DETAILED DESCRIPTION:
BACKGROUND

Since the first case of Severe Acute Respiratory Syndrome - Coronavirus - 2 (SARS-CoV-2) infection and its subsequent clinical manifestation (COronaVIrus Disease 19, COVID-19) in the city of Wuhan (Hubei, China) in December 2019, contagion abruptly spread to different regions of China and, subsequently, to all continents. To date, 1 521 252 cases have been confirmed worldwide. With the first case ascertained in Lombardy at the end of February 2020, Italy soon became the first European country to face the exponential growth in the number of infected people (to date -May 3, 2020-210,717 total cases, currently positive 100,179).The disease turned into an actual health emergency due to the rapid spread and the need of hospitalization and respiratory function support in Intensive Care Unit (ICU) for a significant fraction of the patients. However, the clinical presentation of COVID-19 is non-specific and extremely heterogeneous. Many patients are asymptomatic or exhibit mild symptoms, which include cough, fever, general malaise with myalgias, anosmia and ageusia. The most common changes in blood tests include lymphopenia, thrombocytopenia and increased C-reactive protein and ferritin.

As emerged by clinical data, the viral infection could be divided into three different phases: stage I, asymptomatic incubation period with little or undetectable viral load; stage II, mild symptomatic period with considerable and detectable viral load; stage III, severe symptomatic period with high viral load.

The definitive diagnosis requires a positive molecular test with Real Time PCR (RT-PCR) method for SARS-CoV-2 on nasopharyngeal swab. However, this technique suffers from sub-optimal sensitivity, which may require repetition on bronchoalveolar lavage. The execution of chest CT is therefore essential, as it is characterized by high sensitivity and can detect highly suggestive findings even in patients with negative RT-PCR.

Although the majority of infections resolve spontaneously without the need for specific therapy, up to 20% of patients can develop severe clinical pictures with pneumonia characterized by dyspnea, tachypnea and hypoxemia that requires treatment in a hospital setting. Pulmonary involvement is typically bilateral, peripheral and basal in most cases, presenting on CT scan with multifocal ground glass opacities and interstitial infiltrations; complete resolution usually takes several weeks. Despite active treatment, about 5-10% of cases can precipitate, often suddenly, into critical conditions including respiratory failure, ARDS and multi-organ dysfunction that require ICU admission and are burdened with high mortality.

Even though the understanding of the pathogenesis of COVID-19 is still incomplete, the central role of the immune response in determining the development of severe clinical pictures is increasingly being defined. Organ damage could therefore not be induced by the direct effect of the infection, but mediated by an uncontrolled immune response resulting in the development of a "cytokine storm", as suggested by the high levels of inflammatory cytokines (among which interleukin 6 (IL-6), tumor necrosis factor (TNF) and interferon γ (IFNγ) play a major role) in patients who exhibit severe or fatal disease. To date, no drug has been approved with a specific indication for the treatment of COVID-19. The current treatment encompasses antiviral agents approved for other viral infections, including protease inhibitors (lopinavir and ritonavir), anti-influenza drugs (oseltamivir and arbidol) and compassionate use of nucleotide analogues. Several studies are evaluating the possible effectiveness of the inhibition of pro-inflammatory cytokines activity in preventing or treating severe COVID-19, through the use of immunomodulators (chloroquine and hydroxychloroquine) or monoclonal antibodies such as tocilizumab, which targets the IL-6 receptor. Despite promising preliminary results, a multitude of patients need an immediate treatment while the results of ongoing clinical trials are awaited.

RATIONALE

Although most COVID-19 infections resolve spontaneously without the need for specific therapy, up to 20% of patients can develop severe clinical pictures with interstitial-alveolar pneumonia characterized by dyspnoea, tachypnea and hypoxemia up to an acute respiratory distress syndrome (ARDS), severe respiratory failure and multi-organ dysfunction requiring ICU hospitalization and burdened with high mortality.

To date, the pathogenesis of SARS-CoV-2 pneumonia is poorly understood, but the immune-inflammatory response to infection is progressively emerging as pivotal in the development of severe clinical manifestations. An adequate viral load might stimulate the immune cells to synthesize pro-inflammatory cytokines as interleukin 1 and 6 (IL-1, IL-6), tumor necrosis factor α (TNF α) and attract macrophages, responsible for the secretion of several chemokines that could trigger an unregulated "cytokine storm". A few reports of histological analysis of lung tissue specimens from COVID-19 patients highlighted nonspecific inflammatory changes with the appearance of edema, hyaline membranes and an inflammatory infiltrate dominated mainly by lymphocytes. Peripheral blood tests often reveal lymphocytopenia and a high neutrophil count are found, especially in case of severe disease, with a high value of neutrophil to lymphocyte ratio (NLR), and a relevant increase in circulating pro-inflammatory cytokines levels.

While vaccines and drugs directly targeting the virus are currently being developed and are not yet available, preventing the excessive and uncontrolled cytokine release and inflammatory response could be the key to avoid the occurrence of severe disease.

Different clinical trials are exploring this path, evaluating immunomodulators and monoclonal antibodies targeting mediators such as interleukin 6(IL-6).

Although conventionally fractionated (1.8-2 Gy/fraction) and hypofractionated (> 3 Gy fraction) radiotherapy, used in the field of neoplastic diseases, provides its therapeutic effect also inducing pro-inflammatory molecules, it has widely been documented in the first decades of the last century that low-dose radiotherapy (LD-RT) is potentially effective and relatively safe in the control of acute and/or chronic inflammatory diseases (e.g. skin diseases such as psoriasis, necrotizing abscesses, tendonitis, impingement syndrome).

Many studies reported the effectiveness of radiation treatment after a single application, with a prompt improvement of symptoms, usually occurring within 24 ours and often definitive or long-lasting. Low dose radiotherapy exerts its effect on several cells involved in the immune response: endothelial cells, polymorphonuclear leukocytes, lymphocytes and macrophages. This is true also for pneumonia.

Endothelial cells play a crucial role in the inflammation process, both for the "homing" process of leukocytes, and for the expression of a wide variety of cytokines and growth factors. Different studies have shown that a dose of 0.5 Gy induces an over-expression of tumor growth factor β (TGF-β), which has immunosuppressive activity and leads to a reduction in leukocyte adhesion on endothelial cells.

The leukocyte "rolling" on the endothelium in the sites where inflammation is present represents the initial step of the inflammatory cascade. The effects of LD-RT were analyzed in vitro; after radiation doses of 0.3 - 0.6 Gy, there was a 25-40% reduction in adhesion compared to control after 24 hours from irradiation.

Ionizing radiation at doses below 1 Gy are also capable to polarize macrophages towards the M2 anti-inflammatory phenotype. Conversely, doses greater than 1 Gy tend to induce polarization towards the M1 pro-inflammatory subtype. The use of low doses of radiation seems to act on macrophages also reducing their cytotoxic action, reducing the production of nitric oxide (NO) through to the inhibitory action on the enzyme cytokine inducible nitric oxide synthetase (iNOS) .

Neutrophils play a central role in lung damage induced by Middle East Respiratory Syndrome (MERS) and SARS-CoV, and likewise in COVID-19, as they migrate into the alveoli where they release proteinases and trigger the innate response, with consequent development of cell damage and clinical presentations like ARDs (30,31). Low-dose radiation therapy is able to initiate the apoptotic process of polymorphonuclear granulocytes (neutrophils), thus reducing their cytotoxic activity (32). This treatment can therefore exert an anti-inflammatory activity through several mechanisms of action, with an optimal and long lasting effect demonstrated for a dose of 0.5 Gy (32).

In the absence of a specific treatment, while ongoing trial are evaluating pharmacological approaches and vaccines, innovative approaches could be undertaken to face the emergency and allow a satisfactory management of the disease.

A single fraction radiation treatment delivering low doses to the entire bilateral lung parenchyma (whole lung treatment) is a reasonable and conceptually valid option to inhibit inflammation and obtain a prompt improve of the symptoms in the short term.

Unlike most of the drugs analyzed so far in the framework of COVID-19 infection, low dose radiotherapy is characterized by a minor risk of side effect (negligible, considering the acute phase) and could therefore represent an optimal complementary therapeutic approach due to its safety and absence of interaction with pharmacological treatments. Moreover, this treatment requires less than one hour including treatment planning and administration.

TREATMENT DELIVERY

The patient will undergo radiation treatment on both lungs in a single session. From the physical-dosimetric point of view, the treatment plan will be calculated in an isocentric manner. The isocenter will be positioned at a depth of 10 cm with respect to an anterior skin landmark specifically defined during CT-scan acquisition. The treatment plan will be elaborated using a field in field irradiation technique, with 2 beams each one composed by 3 beamlets: one conformed to the volume resulting by the union of the lungs with a 2 cm margin, the other two will be obtained by shielding the spine and alternately one lung each. This set up allows to obtain a dose distribution in which the vertebral bodies receive a dose lower than 55 cGy with an average lung dose of 70 cGy and maximum lungs dose lower than than 90 centigray (cGy). The Pinnacle ® treatment planning system (TPS) with Collapsed Convolution calculation algorithm will be used. Prescription doses were determined according to data and indications currently published and optimized to minimize the dose to the vertebrae.

ELIGIBILITY:
Inclusion criteria

* Age ≥ 50 years
* Patients with confirmed diagnosis of SARS-Cov2 infection by RT-PCR on nasopharyngeal swab and / or bronchoalveolar lavage (BAL)
* Patient with Brescia Covid Respiratory Severity Scale (BCRSS) score 2-3
* Suggestive picture finding for interstitial pneumonia on chest X-ray and / or chest CT (optional)
* At least 3 of the following laboratory criteria:

  * PCR> 5 times the maximum limit of the normal value
  * Ferritin> 500 ng / ml
  * lactate dehydrogenase (LDH) > 2 times the maximum limit of the normal value
  * D-dimer> 3 times the maximum limit of the normal value
  * Aspartate aminotransferase (AST)> 2 times the maximum limit of the normal value
  * Total lymphocytes <1000 / ml
* Ability to understand and sign informed consent
* Ability to acquire and maintain the set-up necessary for the delivery of radiotherapy treatment
* A negative pregnancy test will be required of patients of childbearing age before starting radiotherapy treatment. Patients with reproductive potential of both sexes will have to agree to use an effective contraceptive method for at least 6 months from the date of treatment.

Exclusion Criteria:

* Age <50 years
* Brescia Covid Respiratory Severity Scale (BCRSS) score greater than 3
* Patients undergoing invasive mechanical ventilation
* Patients with active autoimmune systemic diseases
* Patients with active infections that are not responsive to current treatment
* Patients with a positive pregnancy test
* Impossibility to maintain the set-up necessary for radiotherapy treatment
* Other concomitant treatments for COVID-19 do not represent an exclusion criterion, however they must be reported (specifying the starting date and dosage)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-05-10 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Lenght of hospital stay (days) | Six months
  Evaluation of the feasibility of low-dose radiotherapy treatment of SARS-Cov2 pneumonia, for the purpose of the subsequent implementation of a phase II study; lenght of hospital stay will be recorded
Number of Intensive Care Unit admissions | Six months
  Evaluation of the feasibility of low-dose radiotherapy treatment of SARS-Cov2 pneumonia; the number of intensive care unit admissions will be recorded

SECONDARY OUTCOMES:
Variation of the Brescia COVID-19 Respiratory Severity Scale after treatment | 3, 6 and 10 days
  Variation of the patient's score according to the Brescia COVID-19 Respiratory Severity Scale (minimum value 0, maximum value 8; higher scores mean a worse outcome) with baseline, assessed at 3, 6 and 10 days after treatment.
Occurence of CTCAE 5.0 adverse events | 10 days and 6 months
  Evaluation of the safety and tolerance of the low-dose radiotherapy treatment of SARS-Cov2 ( using the CTCAE 5.0 scale)
Variation of the chest X-ray radiological findings according to Brixia scoring system | 3 and 6 days
  Variation of the radiological findings, assessed by chest X-ray (performed 3 and 6 days after treatment) and defined according to the Brixia scoring system (0-18 scale, with 18 meaning the worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Stefano M Magrini, Prof, Principal Investigator — Brescia University - ASST Spedali Civili Hospital
Locations (1):
- Radiation Oncology Department, ASST SpedaliCivili, Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Yes
All Individual Participant Data that underlie results in the publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available starting six months from the publication and for five years.
Access Criteria: Written request to principal investigator , indicating the details of the data requested, the reasons of the inquiry and the purpose of the data use; data will be released after Local Ethics Committee approval. Data will be released only for no-profit use, in particular for research purposes.